CLINICAL TRIAL: NCT01115543
Title: A Randomized Trial Comparing Pulse Calcitriol and Alfacalcidol for the Treatment of Secondary Hyperparathyroidism in Hemodialysis Patients
Brief Title: Efficacy and Safety of Alfacalcidol Compared to Calcitriol for Treatment of Secondary Hyperparathyroidism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Dr. Kraiwiporn Kiattisunthorn, Siriraj Medical School, Mahidol University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 358/2551
Record Dates: First submitted 2010-05-01; First posted 2010-05-04 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-05

CONDITIONS: Secondary Hyperparathyroidism; End Stage Renal Disease
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Kidney Failure, Chronic | interventions — alfacalcidol; Calcitriol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- calcitriol (Active Comparator): The subjects were randomized to receive calcitriol in a dose-escalating fashion for up to 24 weeks.
  Interventions: Drug: alfacalcidol and calcitriol
- alfacalcidol (Experimental)
  Interventions: Drug: alfacalcidol and calcitriol

INTERVENTIONS:
Drug: alfacalcidol and calcitriol — The initial dose of alfacalcidol was twice that of calcitriol.Both were adjusted to control intact PTH within the ranges of 150-300 pg/ml.

SUMMARY:
This study was performed to determine whether calcitriol provides a therapeutic advantage to alfacalcidol for treatment of secondary hyperparathyroidism in ESRD patients.

DETAILED DESCRIPTION:
Secondary hyperparathyroidism has a significant impact on morbidity and mortality in advanced chronic kidney disease (CKD).Both nonselective and selective vitamin D receptor activators (VDRAs) are demonstrated in many studies for their efficacy on suppression of PTH. Most of them are quite expensive and unavailable in many countries. Calcitriol and alfacalcidol are less expensive and worldwidely distributed. There is only one short-term study which directly compares these two drugs. This study demonstrates that calcitriol is superior to alfacalcidol. However, alfacalcidol is a prohormone of calcitriol. It has to be converted by 25-hydroxylase at the liver to generate 1,25-dihydroxyvitamin D3 to act on target cells. Many pharmacokinetics studies demonstrate that alfacalcidol has lower AUC compared to calcitriol if they are administered in the same dose. Therefore, the authors hypothesize that alfacalcidol may be equivalently efficacious as calcitriol if its dose is adjusted according to the pharmacokinetics studies.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patients who underwent scheduled hemodialysis for at least 3 months with secondary hyperparathyroidism (intact PTH levels > 300 pg/mL)

Exclusion Criteria:

* (1) age < 18 years (2) hypersensitivity to calcitriol or alfacalcidol (3) inadequate dialysis [defined as single-pooled Kt/V (sp-Kt/V) <1.2 and <2.0 for thrice a week and twice a week hemodialysis] (4) corrected serum calcium >10.2 mg/dL or serum phosphate >6 mg/dL after adjusting dialysate calcium and phosphate binders (5) diameter of parathyroid gland >10 mm (6) pregnancy or lactation (7) liver cirrhosis (8) active kidney transplantation (9) previous parathyroidectomy (10) malignancy or chronic infection/inflammation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Reduction of intact parathyroid hormone levels | 48 weeks

SECONDARY OUTCOMES:
hypercalcemia and hyperphosphatemia | 48 weeks
  proportion of the patients who achieved a target PTH, changes in plasma calcium and phosphorus, the proportion of the patients who had hypercalcemia (plasma corrected calcium > 10.8 mg/dl), hyperphosphatemia (plasma phosphorus > 6.0 mg/dl) and calcium-phosphorus products > 55 mg2/dl2 between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Medical School, Bangkok Noi, Bangkok, Thailand